CLINICAL TRIAL: NCT00932373
Title: A Phase I, Open-Label, Dose-Escalation Study of the Safety and Pharmacokinetics of Trastuzumab-MCC-DM1 (PRO132365) Administered Intravenously to Patients With HER2-Positive Metastatic Breast Cancer Who Have Previously Received a Trastuzumab-Containing Regimen
Brief Title: A Study of Trastuzumab-MCC-DM1 Administered Intravenously to Patients With HER2-Positive Metastatic Breast Cancer Who Have Previously Received a Trastuzumab-Containing Regimen
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TDM3569g
Record Dates: First submitted 2009-06-30; First posted 2009-07-03 (Estimated); Results first posted 2015-07-30 (Estimated); Last update posted 2015-08-26 (Estimated); Status verified 2015-08

CONDITIONS: Metastatic Breast Cancer
Keywords: HER2-positive breast cancer; MBC; Trastuzumab emtansine; Herceptin; T-DM1
MeSH Terms: conditions — Breast Neoplasms | interventions — Ado-Trastuzumab Emtansine

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: trastuzumab-MCC-DM1

INTERVENTIONS:
Drug: trastuzumab-MCC-DM1 — Intravenous escalating dose

SUMMARY:
This is a phase I, multicenter, open-label, dose-escalation study of single-agent trastuzumab-MCC-DM1 administered by intravenous (IV) infusion in patients with HER2-positive metastatic breast cancer (MBC) who have previously received trastuzumab. The study will assess the safety, tolerability, and pharmacokinetics of trastuzumab-MCC-DM1 and determine the dose and schedule to be used in Phase II.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented, incurable, locally advanced or metastatic breast cancer
* Evaluable or measurable HER2-positive disease
* History of progression during or within 60 days after treatment with any prior trastuzumab-containing chemotherapy regimen for HER2-positive breast cancer
* Previous treatment with chemotherapy for MBC
* Granulocyte count ≥ 1,500/μL, platelet count ≥ 100,000/μL, and hemoglobin ≥ 9 g/dL
* Serum bilirubin ≤ 1.5 mg/dL; AST, ALT, and alkaline phosphatase ≤ 2.5 × upper limit of normal (ULN) except for: Patients with hepatic metastases: ALT and AST ≤ 5 × ULN Patients with hepatic and/or bone metastases: alkaline phosphatase ≤ 5 × ULN
* Serum creatinine ≤ 1.5 mg/dL or creatinine clearance of ≥ 60 mL/min based on a 24-hour urine collection
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0, 1, or 2
* Women of childbearing potential and men must agree to use an effective method of birth control (e.g., hormonal, barrier) while receiving study treatment

Exclusion Criteria:

* History of significant cardiac disease, unstable angina, CHF, myocardial infarction, or ventricular arrhythmia requiring medication
* History of Grade ≥ 3 hypersensitivity reaction to trastuzumab
* History of any toxicity to trastuzumab that resulted in trastuzumab being permanently discontinued
* Symptomatic brain metastases or any radiation or surgery for brain metastases within 3 months of first study treatment
* Require supplemental oxygen for daily activities
* Grade ≥ 2 peripheral neuropathy
* Bisphosphonate therapy for symptomatic hypercalcemia
* Any chemotherapy, hormonal therapy, radiotherapy, immunotherapy, or biologic therapy for the treatment of breast cancer within 4 weeks of first study treatment
* Any experimental therapy within 4 weeks of first study treatment
* Any major surgical procedure within 4 weeks of first study treatment
* History of clinically symptomatic liver disease, including viral or other hepatitis, current or history of alcoholism, or cirrhosis
* Pregnancy or lactation
* Cardiac troponin I ≥ 0.2 ng/mL
* Ejection fraction < 50% or below the lower limit of normal determined by echocardiogram or MUGA scan
* Prior cumulative doxorubicin dose of > 360 mg/m2 or equivalent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2006-04; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Holden, M.D., Study Director — Genentech, Inc.

REFERENCES:
- [Derived] Beeram M, Krop IE, Burris HA, Girish SR, Yu W, Lu MW, Holden SN, Modi S. A phase 1 study of weekly dosing of trastuzumab emtansine (T-DM1) in patients with advanced human epidermal growth factor 2-positive breast cancer. Cancer. 2012 Dec 1;118(23):5733-40. doi: 10.1002/cncr.27622. Epub 2012 May 30. PMID 22648179

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Approximately four centers in the United States were to participate in the study to enroll approximately 50-60 patients. Between 25 April 2006 and 20 May 2008, 54 patients were enrolled and 52 were treated.
Pre-assignment Details: Two patients enrolled but discontinued the study prior to receiving study treatment drug, thus 52 patients received at least one dose and are included in the baseline and safety analysis data.
Groups:
- Trastuzumab-MCC-DM1 0.3 mg/kg Every 3 Weeks: Trastuzumab-MCC-DM1 0.3 mg/kg administered intravenously (IV) once every 3 weeks
- Trastuzumab-MCC-DM1 0.6 mg/kg Every 3 Weeks: Trastuzumab-MCC-DM1 0.6 mg/kg administered intravenously (IV) once every 3 weeks
- Trastuzumab-MCC-DM1 1.2 mg/kg Every 3 Weeks: Trastuzumab-MCC-DM1 1.2 mg/kg administered intravenously (IV) once every 3 weeks
- Trastuzumab-MCC-DM1 2.4 mg/kg Every 3 Weeks: Trastuzumab-MCC-DM1 2.4 mg/kg administered intravenously (IV) once every 3 weeks
- Trastuzumab-MCC-DM1 3.6 mg/kg Every 3 Weeks: Trastuzumab-MCC-DM1 3.6 mg/kg administered intravenously (IV) once every 3 weeks
- Trastuzumab-MCC-DM1 4.8 mg/kg Every 3 Weeks: Trastuzumab-MCC-DM1 4.8 mg/kg administered intravenously (IV) once every 3 weeks
- Trastuzumab-MCC-DM1 1.2 mg/kg Weekly: Trastuzumab-MCC-DM1 1.2 mg/kg administered intravenously (IV) once a week
- Trastuzumab-MCC-DM1 1.6 mg/kg Weekly: Trastuzumab-MCC-DM1 1.6 mg/kg administered intravenously (IV) once a week
- Trastuzumab-MCC-DM1 2.0 mg/kg Weekly: Trastuzumab-MCC-DM1 2.0 mg/kg administered intravenously (IV) once a week
- Trastuzumab-MCC-DM1 2.4 mg/kg Weekly: Trastuzumab-MCC-DM1 2.4 mg/kg administered intravenously (IV) once a week
- Trastuzumab-MCC-DM1 2.9 mg/kg Weekly: Trastuzumab-MCC-DM1 2.9 mg/kg administered intravenously (IV) once a week
Period: Overall Study
Arm/Group | Trastuzumab-MCC-DM1 0.3 mg/kg Every 3 Weeks | Trastuzumab-MCC-DM1 0.6 mg/kg Every 3 Weeks | Trastuzumab-MCC-DM1 1.2 mg/kg Every 3 Weeks | Trastuzumab-MCC-DM1 2.4 mg/kg Every 3 Weeks | Trastuzumab-MCC-DM1 3.6 mg/kg Every 3 Weeks | Trastuzumab-MCC-DM1 4.8 mg/kg Every 3 Weeks | Trastuzumab-MCC-DM1 1.2 mg/kg Weekly | Trastuzumab-MCC-DM1 1.6 mg/kg Weekly | Trastuzumab-MCC-DM1 2.0 mg/kg Weekly | Trastuzumab-MCC-DM1 2.4 mg/kg Weekly | Trastuzumab-MCC-DM1 2.9 mg/kg Weekly
Started | 3 | 1 | 1 | 1 | 15 | 3 | 3 | 3 | 3 | 16 | 3
Completed | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 1 | 3 | 0
Not Completed | 3 | 1 | 1 | 0 | 14 | 3 | 1 | 3 | 2 | 13 | 3
Not completed — Progressive disease | 3 | 1 | 0 | 0 | 10 | 1 | 0 | 2 | 1 | 9 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 2 | 1
Not completed — Physician Decision | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Dose limiting toxicity | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Clinical progression | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All summaries were based on data from the safety population (patients who received at least one dose of Trastuzumab-MCC-DM1). All summaries were presented for all patients and by dose level and schedule.
Groups:
- Total: Total of all reporting groups
Arm/Group | Trastuzumab-MCC-DM1 0.3 mg/kg Every 3 Weeks | Trastuzumab-MCC-DM1 0.6 mg/kg Every 3 Weeks | Trastuzumab-MCC-DM1 1.2 mg/kg Every 3 Weeks | Trastuzumab-MCC-DM1 2.4 mg/kg Every 3 Weeks | Trastuzumab-MCC-DM1 3.6 mg/kg Every 3 Weeks | Trastuzumab-MCC-DM1 4.8 mg/kg Every 3 Weeks | Trastuzumab-MCC-DM1 1.2 mg/kg Weekly | Trastuzumab-MCC-DM1 1.6 mg/kg Weekly | Trastuzumab-MCC-DM1 2.0 mg/kg Weekly | Trastuzumab-MCC-DM1 2.4 mg/kg Weekly | Trastuzumab-MCC-DM1 2.9 mg/kg Weekly | Total
Number analyzed (Participants) | 3 | 1 | 1 | 1 | 15 | 3 | 3 | 3 | 3 | 16 | 3 | 52
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.7 (10.1) | 47.0 (0) | 61.0 (0) | 58.0 (0) | 52.1 (10.3) | 48.0 (6.0) | 55.3 (10.0) | 53.0 (6.1) | 55.3 (3.2) | 50.9 (14.0) | 58.3 (11.0) | 52.9 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 1 | 1 | 15 | 3 | 3 | 3 | 3 | 16 | 3 | 52
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 1 | 1 | 1 | 15 | 3 | 3 | 3 | 3 | 16 | 3 | 52

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adverse Events (AE), Serious Adverse Events (SAE), AEs With Grade >=3, and AEs Related To Treatment
Description: The time frame for AEs is study treatment initiation until 30 days after last administration of study treatment or at the time of initiation of another anti-cancer therapy, which ever occurs first.
  The time frame for SAEs is study treatment initiation until 90 days after last administration of study treatment or at the time of initiation of another anti-cancer therapy, which ever occurs first.
Time Frame: Study treatment initiation until 30 or 90 days after last administration of study treatment
Population: Safety-evaluable population: All participants who received at least 1 dose of trastuzumab-MCC-DM1
Measure: Number; unit: percentage of participants
Arm/Group | Trastuzumab-MCC-DM1 0.3 mg/kg Every 3 Weeks | Trastuzumab-MCC-DM1 0.6 mg/kg Every 3 Weeks | Trastuzumab-MCC-DM1 1.2 mg/kg Every 3 Weeks | Trastuzumab-MCC-DM1 2.4 mg/kg Every 3 Weeks | Trastuzumab-MCC-DM1 3.6 mg/kg Every 3 Weeks | Trastuzumab-MCC-DM1 4.8 mg/kg Every 3 Weeks | Trastuzumab-MCC-DM1 1.2 mg/kg Weekly | Trastuzumab-MCC-DM1 1.6 mg/kg Weekly | Trastuzumab-MCC-DM1 2.0 mg/kg Weekly | Trastuzumab-MCC-DM1 2.4 mg/kg Weekly | Trastuzumab-MCC-DM1 2.9 mg/kg Weekly
Number analyzed (Participants) | 3 | 1 | 1 | 1 | 15 | 3 | 3 | 3 | 3 | 16 | 3
percentage of participants
  At least 1 AE | 100 | 100 | 100 | 100 | 100 | 100 | 100 | 100 | 100 | 100 | 100
  AEs with Grade >=3 | 33.3 | 100 | 0 | 0 | 46.7 | 100 | 33.3 | 66.7 | 66.7 | 81.3 | 33.3
  At least 1 SAE | 33.3 | 100 | 0 | 0 | 20 | 66.7 | 33.3 | 33.3 | 33.3 | 50 | 0
  AEs related to treatment | 66.7 | 100 | 100 | 100 | 93.3 | 100 | 100 | 66.7 | 100 | 87.5 | 100

2. Secondary Outcome: Percentage of Participants With an Objective Response
Description: The occurrence of an objective response was determined by the investigator according to Response Evaluation Criteria in Solid Tumors (RECIST). An objective response was defined as a complete response or a partial response as determined on 2 consecutive occasions ≥ 4 weeks apart. A complete response was defined as the disappearance of all target lesions or the disappearance of all non-target lesions and normalization of tumor marker level. A partial response was defined as at least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum of the longest diameter of target lesions.
Time Frame: Baseline to the end of the study (up to 3 years 2 months)
Population: Efficacy population: All enrolled participants who received treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Trastuzumab-MCC-DM1 0.3 mg/kg Every 3 Weeks | Trastuzumab-MCC-DM1 0.6 mg/kg Every 3 Weeks | Trastuzumab-MCC-DM1 1.2 mg/kg Every 3 Weeks | Trastuzumab-MCC-DM1 2.4 mg/kg Every 3 Weeks | Trastuzumab-MCC-DM1 3.6 mg/kg Every 3 Weeks | Trastuzumab-MCC-DM1 4.8 mg/kg Every 3 Weeks | Trastuzumab-MCC-DM1 1.2 mg/kg Weekly | Trastuzumab-MCC-DM1 1.6 mg/kg Weekly | Trastuzumab-MCC-DM1 2.0 mg/kg Weekly | Trastuzumab-MCC-DM1 2.4 mg/kg Weekly | Trastuzumab-MCC-DM1 2.9 mg/kg Weekly
Number analyzed (Participants) | 3 | 1 | 1 | 1 | 15 | 3 | 3 | 3 | 3 | 16 | 3
percentage of participants | 0 | 0 | 0 | 100 | 26.7 | 0 | 100 | 66.7 | 66.7 | 37.5 | 0

3. Secondary Outcome: Duration of Objective Response
Description: Duration of objective response was defined as the time from the initial response to disease progression or death from any cause within 30 days of the last dose of trastuzumab emtansine.
Time Frame: Baseline to the end of the study (up to 3 years 2 months)
Population: Efficacy population: All enrolled participants who received treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Trastuzumab-MCC-DM1 2.4 mg/kg Every 3 Weeks | Trastuzumab-MCC-DM1 3.6 mg/kg Every 3 Weeks | Trastuzumab-MCC-DM1 1.2 mg/kg Weekly | Trastuzumab-MCC-DM1 1.6 mg/kg Weekly | Trastuzumab-MCC-DM1 2.0 mg/kg Weekly | Trastuzumab-MCC-DM1 2.4 mg/kg Weekly
Number analyzed (Participants) | 1 | 4 | 3 | 2 | 2 | 6
Months | NA [NA to NA] — Not estimable as the median and/or confidence interval limits were not reached. | 10.5 [4.2 to 10.5] | NA [NA to NA] — Not estimable as the median and/or confidence interval limits were not reached. | 2.9 [NA to NA] — Not estimable as the median and/or confidence interval limits were not reached. | NA [NA to NA] — Not estimable as the median and/or confidence interval limits were not reached. | 5.6 [4.5 to NA] — Not estimable as the median and/or confidence interval limits were not reached.

4. Secondary Outcome: Progression-free Survival
Description: Progression-free survival was defined as the time from first dose of trastuzumab emtansine to documented disease progression or death from any cause within 30 days of the last dose of trastuzumab emtansine, whichever occurred earlier. Progressive disease was defined as at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum of the longest diameter of target lesions recorded since treatment started or the appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions.
Time Frame: Baseline to the end of the study (up to 3 years 2 months)
Population: Efficacy population: All enrolled participants who received treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Trastuzumab-MCC-DM1 0.3 mg/kg Every 3 Weeks | Trastuzumab-MCC-DM1 0.6 mg/kg Every 3 Weeks | Trastuzumab-MCC-DM1 1.2 mg/kg Every 3 Weeks | Trastuzumab-MCC-DM1 2.4 mg/kg Every 3 Weeks | Trastuzumab-MCC-DM1 3.6 mg/kg Every 3 Weeks | Trastuzumab-MCC-DM1 4.8 mg/kg Every 3 Weeks | Trastuzumab-MCC-DM1 1.2 mg/kg Weekly | Trastuzumab-MCC-DM1 1.6 mg/kg Weekly | Trastuzumab-MCC-DM1 2.0 mg/kg Weekly | Trastuzumab-MCC-DM1 2.4 mg/kg Weekly | Trastuzumab-MCC-DM1 2.9 mg/kg Weekly
Number analyzed (Participants) | 3 | 1 | 1 | 1 | 15 | 3 | 3 | 3 | 3 | 16 | 3
Months | 2.7 [1.3 to 4.2] | 1.7 [NA to NA] — Not Estimable | NA [NA to NA] — Not Estimable | NA [NA to NA] — Not Estimable | 10.4 [3.4 to 17.1] | NA [0.7 to NA] — Not Estimable | NA [20.8 to NA] — Not Estimable | 4.5 [1.6 to NA] — Not Estimable | NA [7.2 to NA] — Not Estimable | 5.7 [1.3 to 10.9] | 2.0 [1.3 to 2.8]

5. Secondary Outcome: Percentage of Participants With Anti-therapeutic Antibodies to Trastuzumab Emtansine
Description: After the start of trastuzumab emtansine treatment, serum samples were collected every 3 weeks prior to trastuzumab emtansine dosing for detection of anti-therapeutic antibodies using a validated assay. A bridging antibody electrochemiluminescence assay (ECLA) was used to detect antibodies to trastuzumab emtansine. The assay utilized trastuzumab emtansine conjugated to biotin and a ruthenium label to form a complex with anti-trastuzumab emtansine antibodies. The antibody complex was captured by streptavidin-coated paramagnetic beads.
Time Frame: Baseline to the end of the study (up to 3 years 2 months)
Measure: Number; unit: percentage of participants
Groups:
- Trastuzumab-MCC-DM1 Every 3 Weeks: Trastuzumab-MCC-DM1 0.3 to 4.8 mg/kg administered intravenously (IV) once every 3 weeks
- Trastuzumab-MCC-DM1 Every Weeks: Trastuzumab-MCC-DM1 1.2 to 2.9 mg/kg administered intravenously (IV) once every week
Arm/Group | Trastuzumab-MCC-DM1 Every 3 Weeks | Trastuzumab-MCC-DM1 Every Weeks
Number analyzed (Participants) | 24 | 28
percentage of participants
  Pre-dose (Cycle 1, Day 1) | 0.0 | 3.7
  Any Visit after Dosing | 4.3 | 0.0

6. Primary Outcome: Number of Patients With Dose Limiting Toxicities (DLTs)
Description: DLT is defined as one of the following as per investigator related to study drug:
  * Grade ≥ 3 non-hematologic, non-hepatic major organ toxicity
  * Grade ≥ 3 cardiac toxicity, including cardiac troponin I elevation or any new segmental wall abnormality as determined by non-invasive cardiac imaging
  * Grade ≥ 4 thrombocytopenia
  * Grade ≥ 4 neutropenia (absolute neutrophil count < 500/μ L) lasting > 4 days or accompanied by fever
  * Grade ≥ 4 anemia
  * Grade ≥ 3 serum bilirubin, hepatic transaminase (alanine aminotransferase or aspartate aminotransferase), or alkaline phosphatase For patients with Grade 2 hepatic transaminase or alkaline phosphatase levels at baseline as a result of liver metastases or bone metastases, a hepatic transaminase or alkaline phosphatase level ≥ 10 times the upper limit of normal will be considered a DLT.
  * Weekly cohorts only: Toxicity preventing retreatment on Cycle 1, Day 8 or toxicity preventing re-treatment on Cycle 1, Days 15 and Day 22
Time Frame: A minimum of 21 days after first dose of trastuzumab-MCC-DM1
Population: Safety Population included all treated patients
Measure: Number; unit: participants
Arm/Group | Trastuzumab-MCC-DM1 0.3 mg/kg Every 3 Weeks | Trastuzumab-MCC-DM1 0.6 mg/kg Every 3 Weeks | Trastuzumab-MCC-DM1 1.2 mg/kg Every 3 Weeks | Trastuzumab-MCC-DM1 2.4 mg/kg Every 3 Weeks | Trastuzumab-MCC-DM1 3.6 mg/kg Every 3 Weeks | Trastuzumab-MCC-DM1 4.8 mg/kg Every 3 Weeks | Trastuzumab-MCC-DM1 1.2 mg/kg Weekly | Trastuzumab-MCC-DM1 1.6 mg/kg Weekly | Trastuzumab-MCC-DM1 2.0 mg/kg Weekly | Trastuzumab-MCC-DM1 2.4 mg/kg Weekly | Trastuzumab-MCC-DM1 2.9 mg/kg Weekly
Number analyzed (Participants) | 3 | 1 | 1 | 1 | 15 | 3 | 3 | 3 | 3 | 16 | 3
participants | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 2

7. Primary Outcome: Maximum Tolerated Dose (MTD)
Description: The highest dose level resulting in a DLT in ≤ 1 of 6 patients was declared the MTD.
Time Frame: A minimum of 21 days after first dose of trastuzumab-MCC-DM1
Population: Safety evaluable population: All participants who received at least 1 dose of trastuzumab-MCC-DM1
Measure: Number; unit: mg/kg
Arm/Group | Trastuzumab-MCC-DM1 Every 3 Weeks | Trastuzumab-MCC-DM1 Every Weeks
Number analyzed (Participants) | 24 | 28
mg/kg | 3.6 | 2.4

8. Primary Outcome: Pharmacokinetic (PK) Parameters After the First Dose: Maximum Observed Plasma Concentration Cmax for T-DM1 Concentrations
Time Frame: 3-Week and Weekly Cohorts: Cycle 1 Day 1 Pre-dose 30 minutes and 4 hours after the end of infusion; Cycle 1 Day 2, 3, 4, 8 (Pre-dose 30 minutes after the end of infusion) 11, 15 (Pre-dose 30 minutes after the end of infusion) and 18
Population: Pharmacokinetic-evaluable patients were defined as patients who received at least one dose of T-DM1 with at least one post-dose concentration data point.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Trastuzumab-MCC-DM1 0.3 mg/kg Every 3 Weeks | Trastuzumab-MCC-DM1 0.6 mg/kg Every 3 Weeks | Trastuzumab-MCC-DM1 1.2 mg/kg Every 3 Weeks | Trastuzumab-MCC-DM1 2.4 mg/kg Every 3 Weeks | Trastuzumab-MCC-DM1 3.6 mg/kg Every 3 Weeks | Trastuzumab-MCC-DM1 4.8 mg/kg Every 3 Weeks | Trastuzumab-MCC-DM1 1.2 mg/kg Weekly | Trastuzumab-MCC-DM1 1.6 mg/kg Weekly | Trastuzumab-MCC-DM1 2.0 mg/kg Weekly | Trastuzumab-MCC-DM1 2.4 mg/kg Weekly | Trastuzumab-MCC-DM1 2.9 mg/kg Weekly
Number analyzed (Participants) | 3 | 1 | 1 | 1 | 15 | 3 | 3 | 3 | 3 | 16 | 3
μg/mL | 9.63 (1.73) | 13.3 (0) | 20.3 (0) | 76.3 (0) | 76.2 (19.1) | 130 (7.77) | 29.6 (5.66) | 34.3 (4.81) | 48.0 (9.56) | 54.8 (12.6) | 78.1 (33.9)

9. Primary Outcome: PK Parameters After the First Dose: Area Under the Plasma Concentration-time Curve From 0 to Infinity (AUC[0-∞] for T-DM1 Concentrations
Time Frame: as for outcome 8
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: day • μg/mL
Arm/Group | Trastuzumab-MCC-DM1 0.3 mg/kg Every 3 Weeks | Trastuzumab-MCC-DM1 0.6 mg/kg Every 3 Weeks | Trastuzumab-MCC-DM1 1.2 mg/kg Every 3 Weeks | Trastuzumab-MCC-DM1 2.4 mg/kg Every 3 Weeks | Trastuzumab-MCC-DM1 3.6 mg/kg Every 3 Weeks | Trastuzumab-MCC-DM1 4.8 mg/kg Every 3 Weeks | Trastuzumab-MCC-DM1 1.2 mg/kg Weekly | Trastuzumab-MCC-DM1 1.6 mg/kg Weekly | Trastuzumab-MCC-DM1 2.0 mg/kg Weekly | Trastuzumab-MCC-DM1 2.4 mg/kg Weekly | Trastuzumab-MCC-DM1 2.9 mg/kg Weekly
Number analyzed (Participants) | 3 | 1 | 1 | 1 | 15 | 3 | 3 | 3 | 3 | 16 | 3
day • μg/mL | 14.5 (3.39) | 24.5 (0) | 42.9 (0) | 330 (0) | 300 (65.8) | 673 (12.2) | 76.2 (10.4) | 130 (39.7) | 175 (41.0) | 199 (54.5) | 212 (39.0)

10. Primary Outcome: PK Parameters After the First Dose: Terminal Half-life (t½) for T-DM1 Concentrations
Description: Terminal phase elimination half-life (T1/2) is the time required for half of the drug to be eliminated from the plasma.
Time Frame: as for outcome 8
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: day
Arm/Group | Trastuzumab-MCC-DM1 0.3 mg/kg Every 3 Weeks | Trastuzumab-MCC-DM1 0.6 mg/kg Every 3 Weeks | Trastuzumab-MCC-DM1 1.2 mg/kg Every 3 Weeks | Trastuzumab-MCC-DM1 2.4 mg/kg Every 3 Weeks | Trastuzumab-MCC-DM1 3.6 mg/kg Every 3 Weeks | Trastuzumab-MCC-DM1 4.8 mg/kg Every 3 Weeks | Trastuzumab-MCC-DM1 1.2 mg/kg Weekly | Trastuzumab-MCC-DM1 1.6 mg/kg Weekly | Trastuzumab-MCC-DM1 2.0 mg/kg Weekly | Trastuzumab-MCC-DM1 2.4 mg/kg Weekly | Trastuzumab-MCC-DM1 2.9 mg/kg Weekly
Number analyzed (Participants) | 3 | 1 | 1 | 1 | 15 | 3 | 3 | 3 | 3 | 16 | 3
day | 1.3 (0.2) | 1.3 (0) | 1.3 (0) | 2.2 (0) | 3.1 (0.7) | 4.1 (0.7) | 2.3 (0.6) | 3.4 (0.8) | 3.1 (0.3) | 3.3 (1.1) | 2.9 (0.5)

ADVERSE EVENTS:
Time Frame: Baseline to the end of the study (up to 3 years 2 months)
Groups:
- Trastuzumab-MCC-DM 0.3 mg/kg Every 3 Weeks: Trastuzumab-MCC-DM 0.3 mg/kg administered intravenously (IV) once every 3 weeks
- Trastuzumab-MCC-DM 0.6 mg/kg Every 3 Weeks: Trastuzumab-MCC-DM 0.6 mg/kg administered intravenously (IV) once every 3 weeks
- Trastuzumab-MCC-DM 1.2 mg/kg Every 3 Weeks: Trastuzumab-MCC-DM 1.2 mg/kg administered intravenously (IV) once every 3 weeks
- Trastuzumab-MCC-DM 2.4 mg/kg Every 3 Weeks: Trastuzumab-MCC-DM 2.4 mg/kg administered intravenously (IV) once every 3 weeks
- Trastuzumab-MCC-DM 3.6 mg/kg Every 3 Weeks: Trastuzumab-MCC-DM 3.6 mg/kg administered intravenously (IV) once every 3 weeks
- Trastuzumab-MCC-DM 4.8 mg/kg Every 3 Weeks: Trastuzumab-MCC-DM 4.8 mg/kg administered intravenously (IV) once every 3 weeks
- Trastuzumab-MCC-DM 1.2 mg/kg Weekly: Trastuzumab-MCC-DM 1.2 mg/kg administered intravenously (IV) once a week
- Trastuzumab-MCC-DM 1.6 mg/kg Weekly: Trastuzumab-MCC-DM 1.6 mg/kg administered intravenously (IV) once a week
- Trastuzumab-MCC-DM 2.0 mg/kg Weekly: Trastuzumab-MCC-DM 2.0 mg/kg administered intravenously (IV) once a week
- Trastuzumab-MCC-DM 2.4 mg/kg Weekly: Trastuzumab-MCC-DM 2.4 mg/kg administered intravenously (IV) once a week
- Trastuzumab-MCC-DM 2.9 mg/kg Weekly: 2.9 mg/kg administered intravenously (IV) once a week
Arm/Group | Trastuzumab-MCC-DM 0.3 mg/kg Every 3 Weeks | Trastuzumab-MCC-DM 0.6 mg/kg Every 3 Weeks | Trastuzumab-MCC-DM 1.2 mg/kg Every 3 Weeks | Trastuzumab-MCC-DM 2.4 mg/kg Every 3 Weeks | Trastuzumab-MCC-DM 3.6 mg/kg Every 3 Weeks | Trastuzumab-MCC-DM 4.8 mg/kg Every 3 Weeks | Trastuzumab-MCC-DM 1.2 mg/kg Weekly | Trastuzumab-MCC-DM 1.6 mg/kg Weekly | Trastuzumab-MCC-DM 2.0 mg/kg Weekly | Trastuzumab-MCC-DM 2.4 mg/kg Weekly | Trastuzumab-MCC-DM 2.9 mg/kg Weekly
Serious Adverse Events (participants affected / at risk) | 1/3 | 1/1 | 0/1 | 0/1 | 3/15 | 2/3 | 1/3 | 1/3 | 1/3 | 8/16 | 0/3
Other Adverse Events (participants affected / at risk) | 3/3 | 1/1 | 1/1 | 1/1 | 15/15 | 3/3 | 3/3 | 3/3 | 3/3 | 15/16 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Trastuzumab-MCC-DM 0.3 mg/kg Every 3 Weeks (N=3) | Trastuzumab-MCC-DM 0.6 mg/kg Every 3 Weeks (N=1) | Trastuzumab-MCC-DM 1.2 mg/kg Every 3 Weeks (N=1) | Trastuzumab-MCC-DM 2.4 mg/kg Every 3 Weeks (N=1) | Trastuzumab-MCC-DM 3.6 mg/kg Every 3 Weeks (N=15) | Trastuzumab-MCC-DM 4.8 mg/kg Every 3 Weeks (N=3) | Trastuzumab-MCC-DM 1.2 mg/kg Weekly (N=3) | Trastuzumab-MCC-DM 1.6 mg/kg Weekly (N=3) | Trastuzumab-MCC-DM 2.0 mg/kg Weekly (N=3) | Trastuzumab-MCC-DM 2.4 mg/kg Weekly (N=16) | Trastuzumab-MCC-DM 2.9 mg/kg Weekly (N=3)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Humerus Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Brain Oedema (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral Haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Confusional State (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Trastuzumab-MCC-DM 0.3 mg/kg Every 3 Weeks (N=3) | Trastuzumab-MCC-DM 0.6 mg/kg Every 3 Weeks (N=1) | Trastuzumab-MCC-DM 1.2 mg/kg Every 3 Weeks (N=1) | Trastuzumab-MCC-DM 2.4 mg/kg Every 3 Weeks (N=1) | Trastuzumab-MCC-DM 3.6 mg/kg Every 3 Weeks (N=15) | Trastuzumab-MCC-DM 4.8 mg/kg Every 3 Weeks (N=3) | Trastuzumab-MCC-DM 1.2 mg/kg Weekly (N=3) | Trastuzumab-MCC-DM 1.6 mg/kg Weekly (N=3) | Trastuzumab-MCC-DM 2.0 mg/kg Weekly (N=3) | Trastuzumab-MCC-DM 2.4 mg/kg Weekly (N=16) | Trastuzumab-MCC-DM 2.9 mg/kg Weekly (N=3)
ORAL PAIN (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
ALANINE AMINOTRANSFERASE (Investigations) | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 2 | 0
JOINT SPRAIN (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
DYSPEPSIA (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 0
TUMOUR PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0
URINARY TRACT INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 5 | 1 | 1 | 0 | 0 | 1 | 0
NEPHROLITHIASIS (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 4 | 0 | 1 | 0 | 0 | 9 | 0
NASOPHARYNGITIS (Infections and infestations) | 0 | 0 | 0 | 1 | 3 | 0 | 2 | 0 | 1 | 2 | 0
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 0
VOMITING (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 3 | 0 | 2 | 1 | 0 | 6 | 0
MUCOSAL INFLAMMATION (General disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
PATHOLOGICAL FRACTURE (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
NEUTROPENIA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0
LIPASE INCREASED (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 4 | 1 | 2 | 1 | 1 | 2 | 0
PERIORBITAL OEDEMA (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
TACHYCARDIA (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
OEDEMA PERIPHERAL (General disorders) | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
DIARRHOEA (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 2 | 0 | 3 | 1 | 2 | 6 | 1
NAUSEA (Gastrointestinal disorders) | 2 | 1 | 0 | 1 | 6 | 1 | 3 | 1 | 1 | 7 | 2
WEIGHT DECREASED (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
DISORIENTATION (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 4 | 0 | 1 | 0 | 0 | 0 | 0
DRY SKIN (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 0
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
SYNCOPE (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
TUMOUR NECROSIS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
DRY MOUTH (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 3 | 0 | 1 | 1 | 1 | 7 | 0
IRON DEFICIENCY ANAEMIA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 0
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 3 | 1 | 1 | 0 | 2 | 1 | 1
LACRIMATION INCREASED (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0
DRY EYE (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 3 | 0
RETCHING (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 3 | 0
FLUID RETENTION (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
CHEST PAIN (General disorders) | 1 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 1 | 0
FATIGUE (General disorders) | 1 | 0 | 0 | 1 | 9 | 1 | 3 | 1 | 3 | 10 | 1
FLUSHING (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
TOOTH ABSCESS (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
CHILLS (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 1
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0
INFLUENZA LIKE ILLNESS (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
STOMATITIS (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0
CONSTIPATION (Gastrointestinal disorders) | 2 | 0 | 0 | 1 | 3 | 1 | 1 | 0 | 2 | 4 | 2
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 0 | 0 | 1 | 2 | 2 | 1 | 1 | 2 | 8 | 1
LIVER FUNCTION TEST ABNORMAL (Investigations) | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 1 | 1 | 2 | 1
PYREXIA (General disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 2 | 1 | 2 | 2 | 1
INSOMNIA (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 2 | 3 | 0
MENSTRUAL DISORDER (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
DYSGEUSIA (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 3 | 0
ANAEMIA (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 6 | 0 | 0 | 0 | 1 | 6 | 1
RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
DIZZINESS (Nervous system disorders) | 1 | 0 | 0 | 0 | 2 | 1 | 1 | 1 | 0 | 2 | 0
MENTAL STATUS CHANGES (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
RASH MACULAR (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
ANOREXIA (Metabolism and nutrition disorders) | 2 | 0 | 1 | 0 | 2 | 0 | 2 | 0 | 0 | 4 | 1
DRUG HYPERSENSITIVITY (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
EYE PAIN (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 9 | 3 | 1 | 1 | 2 | 6 | 2
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
NEUROPATHY PERIPHERAL (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 0
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
ASTHENIA (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
CONJUNCTIVITIS (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 0
RALES (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 3 | 1 | 0 | 1 | 2 | 5 | 0
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 4 | 1 | 1 | 1 | 2 | 5 | 0
COLD SWEAT (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
FACIAL PAIN (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
FACE OEDEMA (General disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
VISION BLURRED (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
HEADACHE (Nervous system disorders) | 0 | 0 | 0 | 1 | 5 | 1 | 2 | 1 | 1 | 7 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.